CLINICAL TRIAL: NCT04826874
Title: Affect Labeling - Experimental Evaluation and Behavioral Intervention
Acronym: AL_ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hanna Sahlin, Principal investigator, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-06427
Record Dates: First submitted 2021-03-15; First posted 2021-04-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Emotional Dysregulation
Keywords: Emotional Self-Regulation; Emotion Regulation; Affect labeling; Internet intervention
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: within-individual and randomized control design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Affect Labeling_direct (Experimental): Randomized to immediate two-week, internet delivered psychoeducative course in affect labeling
  Interventions: Behavioral: Affect labeling
- Wait-list (No Intervention): Randomized to a two-week wait-list control

INTERVENTIONS:
Behavioral: Affect labeling — Short behavioral intervention teaching affect labeling
  Arms: Affect Labeling_direct

SUMMARY:
The overall aim of this project is to better understand the emotion regulating effect of labeling emotions (affecting labeling, AL) for individuals with self-perceived emotional regulation difficulties from both a clinical population and a non-clinical population, by using both self-assessment and psychophysiological testing of emotional activation. The main part of the project includes a brief intervention aiming to test the emotion-regulating effect of a short behavioral intervention to learn and practice AL. This two-week intervention, aims to improve the ability to regulate emotions, and to assess the benefits of emotion regulation strategies for individuals with and without a clinical diagnosis, but with self-perceived difficulties in emotion regulation.

The second part of this study aims to conceptually replicate a previous basic research study on AL and its emotion-regulating effect in a experimental laboratory setting and to extend that replication to include a clinical group. The replication contributes to an indepth understanding of AL as an implicit emotion regulation strategy in the short term, i.e. as a strategy used directly in the emotionally charged situation, and expands that knowledge to also include the effect in individuals with a clinical diagnosis. Also, it provides the opportunity to evaluate the effect of the two week AL behavioral intervention using psychophysiological testing.

DETAILED DESCRIPTION:
Main study: AFFECT LABELING - DAILY EXERCISE IN PUTTING WORDS ON EMOTIONS DESIGN AND PROCEDURE This clinical study is a randomized, wait-list controlled design with repeated measurements. Participants are randomized at inclusion between being directly offered a 14-day course to train AL and waiting two weeks before beginning the intervention. Participants are blind to this randomization and do not know that they are in the waitlist condition, in order to avoid nocebo effects. The randomization is done 1: 1, and stratified by clinical categorization (participants with or without a psychiatric diagnosis).

The course is given via a secure web platform (BASS4) in which the participant also makes all their assessments, and interacts with the study material and their course leader (clinical psychologist or master level psychology students).

Intervention - web course in affect labeling The intervention is given as a two week internet-delivered course in using AL with the guidance of a course leader (licensed psychologist or psychologist assistant under supervision). The course is divided into two modules where module 1 contains a) Psychoeducation about different emotions and its function, b) Information about AL and its potential emotion-regulating effect, c) Instruction on how to use AL in everyday life and d) Planning of daily short exercises in naming emotions. Daily registration with multiple choice answers is introduced to help the practice of AL. All assessments are web-based and reminders are sent to the participants' cellphone. The course leader is active in providing feedback on the exercises and planning.

Module 2 is largely a continuation of module 1 where any obstacles and other difficulties are discussed in order to increase the chance of active practice in AL, and continued daily practice. Module 3 is a brief summary of what has been taught and is made available to the participant after post-assessment.

Laboratory sub-study: Participants will also participate in a laboratory-based study where the emotion regulating effect of AL will be compared with distraction or passive viewing while being exposed to emotionally provocative visual stimuli. Participants are exposed to 3 blocks of 8 images and questions about the images ("trials") with equal numbers of negative and neutral valence in three conditions: instruction to "Watch", instruction to use AL and instruction to use Distraction. The instructions and pictures are given in a randomized, balanced order. Before each block, a 3-second instruction is displayed that indicates whether the participant should use "Watch", "AL" or "Distraction" for all 8 images in the block.

All participants will carry out the laboratory sub-study on two occasions: before and after the 14 day period it takes for the individuals who directly receives the web-based course in AL to complete it.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient skills in Swedish to be able to fill in self-assessment questionnaires.
* State at least a 3 (or higher) out of 10 regarding everyday difficulties with emotion regulation according to a scale created for this purpose: Do you feel that you currently have problems regulating your emotions? Circle the number that is best for you "(0 no problems at all, 10 Very severe problems.
* Answer "Yes, very much" or "Yes" to the following question: "Would you like to learn to regulate/manage your emotions better?" with the options "Yes, very much / Yes / Maybe, but doubtful if it is worth the effort, does not fit right now / No".

Exclusion Criteria:

* Psychiatric or somatic status that may prevent the participant from completing the experiment or require some form of care intervention the participant does not already undergo.
* Medium to high risk of suicide.
* Moderate to severe self-harming behavior.
* Blood phobia.
* Regular medication with benzodiazepines (including sleep medication, ex Stilnoct).
* Ongoing treatment with emotion regulation elements.

To be part of the clinical group, the participant must state a diagnosis established by a medical professional in the last 5 years, which involves clinical difficulties with emotion regulation such as binge eating disorder, emotional instability, generalized anxiety, depression, social anxiety or ADHD, and does not plan to start, change or discontinue any psychosocial or pharmacological treatment within the next 4 weeks. The non-clinical group must not have been diagnosed or treated for mental illness in the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in The Difficulties in Emotion Regulation Scale, DERS (Gratz & Roemer, 2004) | At day 1 and at day 14 (+/- 5 days)
  Min 36, Max 180. Higher scores represents worse outcome

SECONDARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | At baseline and day 14 (+/- 5 days)
  Min 0, Max 27. Higher scores represents worse outcome
The Generalized Anxiety Disorder 7-item Scale (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006). | At baseline and day 14 (+/- 5 days)
  Min 0, Max 21. Higher scores represents worse outcome
The Emotion Regulation Questionnaire (ERQ; Gross & John, 2003) | At day 1 and day 14 (+/- 5 days)
  Two sub scales: Cognitive reappraisal: Min 6 Max 42. Higher scores represents higher use of reappraisal. Suppression: Min 4 Max 28. Higher scores represents more use of suppression.
The Toronto Alexithymia Scale (TAS-20; Bagby et al., 1994). | At baseline and day 14 (+/- 5 days)
  Min 20, Max 100. Higher scores represents worse outcome
The Ruminative responses scale - Brooding and Reflection (RRS-BR; Treynor et al., 2003, Cronwall, 2019). | At baseline and day 14 (+/- 5 days)
  Min 10 Max 40. Higher scores represents worse outcome
the Client Satisfaction Questionnaire, 8 item (CSQ-8; Attkisson & Zwick, 1982). | At day 14 (+/- 5 days)
  Min 8 Max 32 Higher scores represents better outcome
Levels of expected emotional upset | At day 1 and day 14 (+/- 5 days)
  9-degree Likert scale. Min 1 (Not upset at all) Max 9 (Very upset).
Change in skin conductance response between three different emotion regulation conditions | 3*8*5 seconds at Day 1 and at Day 14 (+/-5 days)
  changes in skin conductance, mean (micro-Siemens (μS)) between the different emotion regulation conditions
Change in Heart Rate Variability (HRV) (micro-Siemens (μS)) averaged over a 5 sec time window, and repeated 8 times per condition, ie. 8*5 seconds repeated 3 times. | At day 1 and at day 14 (+/- 5 days)
  Heart Rate Variability is a measure which indicates the variation in your heartbeats within a specific timeframe.
Change in The Affect Labeling Questionnaire, ALQ (Sahi, et al. (in prep) | At day 1 and at day 14 (+/- 5 days)
  Min 12, Max 60. Higher scores represents better outcome
Change in Experienced emotional upset (Time frame: averaged over a 5 sec time window, repeated 24 times during the experiment) | At day 1 and day 14 (+/- 5 days)
  9-degree Likert scale. Min 1 (Not upset at all) Max 9 (Very upset).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sahlin, Med Dr, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, department of clinical neuroscience, Stockholm, Stockholm County, Sweden